CLINICAL TRIAL: NCT01713595
Title: Inhaled Hypertonic Saline for the Treatment of Acute Lung Injury
Brief Title: Safety Study of Inhaled Saline in Acute Lung Injury
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: difficult getting subjects
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Richard A. Oeckler, M.D., Ph.D., Assistant Professor of Medicine and Physiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-001723
Record Dates: First submitted 2012-10-04; First posted 2012-10-25 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Edema
Keywords: Acute Lung Injury; Mechanical Ventilation
MeSH Terms: conditions — Pulmonary Edema; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypertonic Saline Aerosol (Experimental): a single 5ml dose of 7% Saline aerosol
  Interventions: Drug: Hypertonic Saline Aerosol

INTERVENTIONS:
Drug: Hypertonic Saline Aerosol — A single 5ml dose of 7% Saline aerosol
  Other Names: Nebulized hypertonic saline

SUMMARY:
To determine if an inhaled hypertonic saline solution has any effect on lung function in patients with acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
Hypertonic Saline (HS) aerosols have proven efficacious mucolytics in patient with cystic fibrosis and are well tolerated in that population. Safety concerns in mechanically ventilated patients with ARDS center primarily on HS's effects on lung water distribution (intra vs. extra alveolar) and on airway reactivity. For that reason we plan a small feasibility trial with narrowly focused physiologic endpoints, namely to measure the effects of a single 5ml dose of 7% Saline aerosol on blood gas tensions, hemodynamics and the static and dynamic properties of the relaxed respiratory system. This narrowly scoped study is to lay the foundation for a larger multicenter intervention trial.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will include consenting adult patients (age > 18), who had been intubated and mechanically ventilated for <72 hours and meet international consensus criteria for ARDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Dynamic Compliance of the Respiratory System | Between 5 & 10 minutes before aerosol delivery and 5 to 10 minutes after completion of the aerosol delivery
  Changes in the static and dynamic properties of the respiratory system are surrogate markers of a change in airway tone and/or of the amount and distribution of alveolar edema

SECONDARY OUTCOMES:
Patient-Ventilator Interactions | 5 minutes before aersosol delivery, during the 15 minutes while aerosol is being delivered and 5 minutes after completion of the aerosol delivery
  "Fighting" the ventilator may reflect irritant receptor feedback and related dyspnea and will speak to the feasibility/patient acceptance of the proposed therapy

OTHER OUTCOMES:
Arterial Blood Gas Tension | Between 5 & 10 minutes before aerosol delivery and 5 to 10 minutes after completion of the aerosol delivery
  Changes in oxygenation and CO2 elimination reflect changes in ventilation-perfusion distribution secondary to changes in bronchomotor tone and/or lung water.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Oeckler, M.D., Ph.D., Principal Investigator — Mayo Clinic